CLINICAL TRIAL: NCT02011269
Title: A Randomized, Blinded, Placebo-controlled Multicenter Study to Assess the Safety and Efficacy of Trichuris Suis Ova for the Treatment of Moderate to Severe Chronic Plaque Psoriasis
Brief Title: TSO for Plaque Psoriasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not conducted
Sponsor: Coronado Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNDO 201-201; CNDO 201-201 (Other: Coronado Biosciences)
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Plaque Psoriasis
Keywords: TSO; Ova; Psoriasis; plaque psoriasis; plaque-type; Coronado; Moderate to severe plaque psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 7500 TSO (Active Comparator): 7500 active Trichuris suis ova will be provided in a15 mL of aqueous suspension (supplied in 30 mL glass containers) administered orally, once every 2 weeks for 10 weeks
  Interventions: Biological: Trichuris Suis Ova
- 15000 TSO (Active Comparator): 15000 active Trichuris suis ova will be provided in two 15 mL of aqueous suspension (supplied in 30 mL glass containers) administered orally, once every 2 weeks for 10 weeks
  Interventions: Biological: Trichuris Suis Ova
- Non-active treatment (Placebo Comparator): The TSO placebo drug product is a non-sterile, 15 mL aqueous solution containing phosphate buffer, pH 5 and 0.05% potassium sorbate as antimicrobial preservative. The TSO placebo is supplied in two 30 mL glass containers that is identical to the container/closure described above for the active drug product.
  Interventions: Biological: Trichuris Suis Ova

INTERVENTIONS:
Biological: Trichuris Suis Ova
  Other Names: TSO

SUMMARY:
This is a randomized, blinded, multicenter study to assess the safety and treatment effect of 12 weeks of Trichuris suis ova in subjects diagnosed with moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 to 75 years old.
* Diagnosis of stable plaque type psoriasis for at least 6 months prior to baseline
* Baseline moderate to severe psoriasis, defined as both of the following:

  1. Psoriasis covering a body surface area (BSA) ≥ 10%, and;
  2. PGA ≥ 3, and;
  3. PASI ≥ 12

Exclusion Criteria:

* Patients who are currently taking or have taken in the past 30 days, for any reason, any medication that, in the opinion of the investigator, suppressed the immune response. This may include but is not limited to systemic steroids, azathioprine, methotrexate, cyclosporine, FK506, mycophenolate mofetil, mycophenolic acid, etanercept, adalimumab, infliximab, ustekinumab, cimzia, or any other biologic agent targeted to any cell or cytokine in the immune system. Patients who are on inhaled or ophthalmic steroids are allowed.
* Patients who have demonstrated a primary lack of response to any one of the following biologic agents: etanercept, adalimumab, infliximab or ustekinumab. Patients who initially responded to one of these agents but subsequently lost response (secondary lack of response) are eligible for study entry; however, secondary lack of response to more than one of these agents will exclude the patient from study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Mean percent change in Psoriasis Area and Severity Index (PASI) score | 12 weeks
  Mean percent change in Psoriasis Area and Severity Index (PASI) score from pre-treatment at Week 0 to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ryan, Study Director — Coronado Biosciences